CLINICAL TRIAL: NCT02397213
Title: Ciclosporin to Protect Renal Function In Cardiac Surgery: CiPRICS A Phase II Double Blind Randomized Placebo Controlled Study
Brief Title: Ciclosporin to Protect Renal Function In Cardiac Surgery
Acronym: CiPRICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: NeuroVive Pharmaceutical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014-004610-29
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Acute Kidney Injury
Keywords: Ciclosporin; Acute Kidney injury; Cardiac surgery; Ischemia; Safety; Cystatin C
MeSH Terms: conditions — Acute Kidney Injury; Ischemia | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): All components of the CicloMulsion® emulsion except ciclosporin: soybean oil (refined), triglycerides (medium-chain), egg lecithin, glycerol, oleic acid, sodium hydroxide and water for injection (=0.5 ml/kg).
  Interventions: Drug: Placebo
- Ciclosporin (Active Comparator): Single dose of CicloMulsion® 5 mg/ml, 2.5 mg/kg (=0.5 ml/kg) as intravenous injection.
  Interventions: Drug: Ciclosporin

INTERVENTIONS:
Drug: Ciclosporin — Single dose of CicloMulsion® 5 mg/ml, 2.5 mg/kg (=0.5 ml/kg) as intravenous injection preoperatively after anesthesia induction.
  Other Names: CicloMulsion® ATC-code: CO1EB
  Arms: Ciclosporin
Drug: Placebo — All components of the CicloMulsion® emulsion except ciclosporin: soybean oil (refined), triglycerides (medium-chain), egg lecithin, glycerol, oleic acid, sodium hydroxide and water for injection (=0.5 ml/kg).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the potential of ciclosporin in reducing risk and degree of acute kidney injury after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication after cardiac surgery and is associated with decreased long-term survival. The mechanism for inducing acute kidney injury is unknown but ischaemia-reperfusion injury is indicated to be a part of the cause.

Animal studies have showed cytoprotective, preconditioning and anti-apoptotic effects of ciclosporin in ischaemia-reperfusion injury in the kidney. The major mechanism is thought to be inhibition of the reperfusion triggered opening of the mitochondrial permeability transition pore (mPTP), responsible for reperfusion-induced necrosis. During cardiac surgery, the period of extracorporeal circulation (ECC) changes the perfusion through the kidney. Return to normal perfusion with a beating heart has similarities with reperfusion following ischemia.

Administration of ciclosporin in conjunction with percutaneous coronary intervention (PCI), heart surgery and traumatic brain injury (TBI) in humans has shown to be safe with no direct side-effects.

The investigators therefore hypothesize that a preconditioning effect of ciclosporin before coronary artery bypass grafting (CABG) can reduce the level of renal dysfunction after this type of cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent CABG
* Written informed consent to participate
* Preoperative CyC eGFR or MDRD eGFR is 90-15.

Exclusion Criteria:

* Uncontrolled hypertension
* Hypersensitivity to ciclosporin or any of the excipients of the lipid emulsion, including egg-, soya- or peanut protein
* Pregnancy or fertile woman
* Ciclosporin treatment within 4 weeks
* Ongoing malignancy, ongoing immunosuppressive treatment, severe hepatic dysfunction, dialysis or severe infection
* Ongoing medication with dabigatran, aliskiren, bosentan, stiripentol, glibenclamid, St John's worth, or
* Off-pump surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ciclosporin to Protect Renal function In Cardiac Surgery. | up to day 3
  Relative P-CyC change from day -1 to day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Bjursten, Md, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skane University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Ederoth P, Grins E, Dardashti A, Bronden B, Metzsch C, Erdling A, Nozohoor S, Mokhtari A, Hansson MJ, Elmer E, Algotsson L, Jovinge S, Bjursten H. Ciclosporin to Protect Renal function In Cardiac Surgery (CiPRICS): a study protocol for a double-blind, randomised, placebo-controlled, proof-of-concept study. BMJ Open. 2016 Dec 15;6(12):e012299. doi: 10.1136/bmjopen-2016-012299. PMID 27979834